CLINICAL TRIAL: NCT00721734
Title: Phase 2 Study of the Safety and Pharmacokinetics of Carfilzomib in Subjects With Relapsed and Refractory Multiple Myeloma and Varying Degrees of Renal Function
Brief Title: Study of the Safety and Pharmacokinetics of Carfilzomib in Patients With Relapsed and Refractory Multiple Myeloma and Varying Degrees of Renal Function
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PX-171-005
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Results first posted 2015-12-09 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Multiple Myeloma; Renal Insufficiency
Keywords: Myeloma; Renal Insufficiency; Proteasome; Hematological; carfilzomib; PR-171
MeSH Terms: conditions — Multiple Myeloma; Renal Insufficiency; Neoplasms, Plasma Cell | interventions — carfilzomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Carfilzomib (Experimental): Carfilzomib, 15 mg/m², was administered intravenously (IV) on Days 1, 2, 8, 9, 15, and 16 of repeated 28-day cycles for a maximum of 12 cycles.
  If the 15 mg/m² dose was tolerated the dose could be increased to 20 mg/m² starting at Cycle 2. If 20 mg/m² was tolerated, an additional dose escalation to 27 mg/m² was allowed at Cycle 3 or at subsequent cycles.
  Interventions: Drug: Carfilzomib

INTERVENTIONS:
Drug: Carfilzomib — Carfilzomib was administered intravenously (IV) at a rate of approximately 10 mL/minute.
  Other Names: PR-171; Kyprolis®

SUMMARY:
The purpose of this study is to assess the influence of renal impairment on carfilzomib in patients with Multiple Myeloma (MM).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent in accordance with federal, local, and institutional guidelines
2. Males and females ≥ 18 years of age
3. Multiple Myeloma
4. Documented relapsed or progressive disease (PD) after receiving at least two prior treatment regimens (induction therapy with autologous stem cell transplant and maintenance is considered a single regimen), and must have achieved a minimal response or better to at least one of the regimens
5. Current measurable disease, as indicated by one or more of the following:

   * Serum M-protein ≥ 0.5 g/dL
   * Urine M-protein ≥ 200 mg/24 hours
   * Serum Free Light Chain (FLC) assay: Involved FLC level ≥ 10 mg/dL provided serum FLC ratio is abnormal
6. Life expectancy of more than three months
7. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
8. Adequate hepatic function, with bilirubin < 2 times the upper limit of normal (ULN) and alanine aminotransferase (ALT) < 3 times ULN
9. Total white blood cell (WBC) count ≥ 2,000/mm³
10. Absolute neutrophil count (ANC) ≥ 1,000/mm³
11. Hemoglobin ≥ 7 gm/dL

    * Subjects may receive red blood cell (RBC) transfusions or supportive care with erythropoietin or darbepoetin in accordance with institutional guidelines
12. Platelet count ≥ 30,000/ mm³
13. Female subjects of child-bearing potential must have a negative serum pregnancy test within seven days of the first dose and agree to use dual methods of contraception during and for 3 months following last dose of drug. Post menopausal females (> 45 years old and without menses for > 1 year) and surgically sterilized females are exempt from a pregnancy test
14. Male subjects must use an effective barrier method of contraception during study and for three months following the last dose if sexually active with a female of child-bearing potential

Exclusion Criteria:

1. Glucocorticoid therapy in a dose equivalent to prednisone ≥ 20 mg/day within 14 days prior to first dose of study drug
2. POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
3. Plasma cell leukemia
4. Chemotherapy with approved or investigative anticancer therapeutics, including steroid therapy dose as defined above, within 14 days prior to first dose of study drug or antibody therapy within 6 weeks prior to first dose of study drug
5. Radiation therapy or immunotherapy within 3 weeks prior to first dose; localized radiation therapy within 1 week prior to first dose
6. Participation in an investigational therapeutic study within 14 days prior to first dose of study drug
7. Prior carfilzomib treatment
8. Pregnant or lactating females
9. Major surgery within 3 weeks prior to first dose of study drug
10. Congestive heart failure (New York Heart Association Class III to IV), symptomatic ischemia, conduction abnormalities or myocardial infarction in the three months prior to first dose of study drug
11. Uncontrolled hypertension
12. Recent history of acute active infection requiring systemic antibiotics, antivirals, or antifungals within two weeks prior to first dose of study drug
13. Known or suspected human immunodeficiency virus (HIV) infection, known HIV seropositivity
14. Active hepatitis A, B, or C infection
15. Other malignancy within the past 3 years except a) adequately treated basal cell or squamous cell skin cancer, b) carcinoma in situ of the cervix, or c) prostate cancer < Gleason Grade 7 with stable prostate specific antigen (PSA) levels
16. Any clinically significant medical or psychiatric disease or condition that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent
17. Significant neuropathy (Grade 3, Grade 4, or Grade 2 with pain) at the time of the first dose and/or within 14 days prior to enrollment
18. Subjects in whom the required program of oral hydration and intravenous fluid hydration is contraindicated, e.g., due to preexisting pulmonary or cardiac impairment
19. Subjects with pleural effusions requiring routine thoracentesis or ascites requiring routine paracentesis
20. Subjects with a known contraindication to receiving dexamethasone or allopurinol
21. Receipt of granulocyte- and granulocyte/ macrophage- colony stimulating factor (G-CSF and GM-CSF) within 1 week prior to first dose of study drug
22. Receipt of pegylated G-CSF within 2 weeks prior to first dose of study drug
23. RBC and platelet transfusions within 7 days prior to first dose of study drug
24. Subjects with known or suspected cardiac amyloidosis
25. Subjects with myelodysplastic syndrome
26. Subjects undergoing peritoneal dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (5):
- United States (5):
  - University of California- San Francisco, San Francisco, California
  - University of Maryland Medical Center, Baltimore, Maryland
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Cornell University, New York, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled patients with multiple myeloma (MM) who had relapsed or progressive disease (PD) after at least 1 (original protocol) or 2 (following protocol Amendment 1) prior therapeutic treatments or regimens. Five groups of MM patients, representing different levels of renal function, were evaluated.
Groups:
- Carfilzomib - Normal RF: Participants with normal renal function (RF; defined as 24-hour urine creatinine clearance (CrCL) > 80 mL/minute) received carfilzomib, 15 mg/m², administered intravenously (IV) on Days 1, 2, 8, 9, 15, and 16 of repeated 28-day cycles for a maximum of 12 cycles.
  If the 15 mg/m² dose was tolerated the dose could be increased to 20 mg/m² starting at Cycle 2. If 20 mg/m² was tolerated, an additional dose escalation to 27 mg/m² was allowed at Cycle 3 or at subsequent cycles.
- Carfilzomib - Mild RI: Participants with mild renal impairment (RI; CrCL between 50-80 mL/minute) received carfilzomib, 15 mg/m², administered intravenously on Days 1, 2, 8, 9, 15, and 16 of repeated 28-day cycles for a maximum of 12 cycles.
  If the 15 mg/m² dose was tolerated the dose could be increased to 20 mg/m² starting at Cycle 2. If 20 mg/m² was tolerated, an additional dose escalation to 27 mg/m² was allowed at Cycle 3 or at subsequent cycles.
- Carfilzomib - Moderate RI: Participants with moderate renal impairment (CrCL between 30-49 mL/minute) received carfilzomib, 15 mg/m², administered intravenously on Days 1, 2, 8, 9, 15, and 16 of repeated 28-day cycles for a maximum of 12 cycles.
  If the 15 mg/m² dose was tolerated the dose could be increased to 20 mg/m² starting at Cycle 2. If 20 mg/m² was tolerated, an additional dose escalation to 27 mg/m² was allowed at Cycle 3 or at subsequent cycles.
- Carfilzomib - Severe RI: Participants with severe renal impairment (CrCL < 30 mL/minute) received carfilzomib, 15 mg/m², administered intravenously on Days 1, 2, 8, 9, 15, and 16 of repeated 28-day cycles for a maximum of 12 cycles.
  If the 15 mg/m² dose was tolerated the dose could be increased to 20 mg/m² starting at Cycle 2. If 20 mg/m² was tolerated, an additional dose escalation to 27 mg/m² was allowed at Cycle 3 or at subsequent cycles.
- Carfilzomib - Dialysis: Participants undergoing chronic hemodialysis received carfilzomib, 15 mg/m², administered intravenously on Days 1, 2, 8, 9, 15, and 16 of repeated 28-day cycles for a maximum of 12 cycles.
  If the 15 mg/m² dose was tolerated the dose could be increased to 20 mg/m² starting at Cycle 2. If 20 mg/m² was tolerated, an additional dose escalation to 27 mg/m² was allowed at Cycle 3 or at subsequent cycles.
Period: Overall Study
Arm/Group | Carfilzomib - Normal RF | Carfilzomib - Mild RI | Carfilzomib - Moderate RI | Carfilzomib - Severe RI | Carfilzomib - Dialysis
Started | 12 | 12 | 10 | 8 | 8
Completed | 4 (Completed 12 cycles of carfilzomib treatment) | 0 (Completed 12 cycles of carfilzomib treatment) | 2 (Completed 12 cycles of carfilzomib treatment) | 2 (Completed 12 cycles of carfilzomib treatment) | 2 (Completed 12 cycles of carfilzomib treatment)
Not Completed | 8 | 12 | 8 | 6 | 6
Not completed — Progressive Disease | 3 | 10 | 4 | 5 | 2
Not completed — Adverse Event | 3 | 1 | 4 | 0 | 3
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carfilzomib - Normal RF | Carfilzomib - Mild RI | Carfilzomib - Moderate RI | Carfilzomib - Severe RI | Carfilzomib - Dialysis | Total
Number analyzed (Participants) | 12 | 12 | 10 | 8 | 8 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 8 | 4 | 1 | 7 | 26
  >=65 years | 6 | 4 | 6 | 7 | 1 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (5.70) | 63.5 (7.85) | 66.2 (9.65) | 73.0 (8.23) | 56.0 (7.91) | 64.6 (9.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 3 | 3 | 4 | 22
  Male | 8 | 4 | 7 | 5 | 4 | 28
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 2 | 2 | 4 | 1 | 2 | 11
  Asian/Pacific Islander | 0 | 2 | 0 | 0 | 1 | 3
  Caucasian | 10 | 8 | 6 | 7 | 5 | 36
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is used by doctors and researchers to assess how a participants disease is progressing, assess how the disease affects the daily living activities of the participant and determine appropriate treatment and prognosis. 0 = Fully Active; 1 = Restricted activity but ambulatory; 2 = Ambulatory but unable to carry out work activities; 3 = Limited Self-Care; 4 = Completely Disabled, no self-care, confined to bed or chair; 5 = Dead.
  participants
    0 (Fully active) | 4 | 2 | 0 | 2 | 0 | 8
    1 (Restrictive but ambulatory) | 8 | 9 | 9 | 1 | 5 | 32
    2 (Ambulatory but unable to work) | 0 | 1 | 1 | 5 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Clearance (CL) of Carfilzomib on Day 1 of Cycle 1
Description: Plasma concentrations of carfilzomib was determined by a validated liquid chromatography tandem mass spectrometry (LC MS/MS) method. The lower limit of quantitation (LLOQ) was 0.300 ng/mL. Concentration values that were below the LLOQ (BLQ) were set to zero. Pharmacokinetic (PK) parameters were calculated from the individual plasma concentrations of carfilzomib using a noncompartmental method.
Time Frame: Cycle 1, Day 1 before dosing, at the end of the injection, 5, 15, 30, and 60 minutes, and 1.5, 2, 4, 6 and 24 hours postdose.
Population: The pharmacokinetic (PK) evaluable population includes participants with stable baseline renal function (Arms 1-4) who completed all protocol-specified treatment and PK blood sample collection through Cycle 1, Day 16. In Group 5, only samples collected before dialysis were included.
  CL could not be estimated for 11 patients in the PK population.
Measure: Mean (Standard Deviation); unit: liters/hour
Arm/Group | Carfilzomib - Normal RF | Carfilzomib - Mild RI | Carfilzomib - Moderate RI | Carfilzomib - Severe RI | Carfilzomib - Dialysis
Number analyzed (Participants) | 6 | 6 | 3 | 4 | 5
liters/hour | 151 (79.3) | 113 (40.7) | 288 (264) | 170 (58.4) | 170 (60.2)
Statistical Analysis 1: Comparison: Carfilzomib - Normal RF vs Carfilzomib - Mild RI vs Carfilzomib - Moderate RI vs Carfilzomib - Severe RI; In order to estimate a possible effect of renal function, the relationship between the clearance of carfilzomib and creatinine clearance (CrCl) was explored using a mixed-effects model that included CrCl. The slope of the regression of CL as a function of CrCL at Cycle 1, Day 1 was evaluated using a linear regression model that included CrCL as continuous variables (excluding the hemodialysis group); Test type: Superiority or Other; p = 0.4114, Regression, Linear; Slope = -0.607, 95% CI 2-sided [-2.129 to 0.914]

2. Secondary Outcome: Clearance (CL) of Carfilzomib on Day 15 of Cycle 1
Time Frame: Cycle 1, Day 15 before dosing, at the end of the injection, 5, 15, 30, and 60 minutes, and 1.5, 2, 4, 6 and 24 hours postdose.
Population: The pharmacokinetic (PK) evaluable population with available data
Measure: Mean (Standard Deviation); unit: liters/hour
Arm/Group | Carfilzomib - Normal RF | Carfilzomib - Mild RI | Carfilzomib - Moderate RI | Carfilzomib - Severe RI | Carfilzomib - Dialysis
Number analyzed (Participants) | 5 | 5 | 3 | 1 | 5
liters/hour | 660 (1134) | 115 (34.7) | 119 (16.5) | 110 (NA) — Can not be calculated for a sample of 1 | 114 (61.2)

3. Secondary Outcome: Clearance (CL) of Carfilzomib on Day 15 of Cycle 2
Time Frame: Cycle 2, Day 15, before dosing, at the end of the injection, 5, 15, 30, and 60 minutes, and 1.5, 2, 4, 6 and 24 hours postdose.
Population: The pharmacokinetic (PK) evaluable population with available data
Measure: Mean (Standard Deviation); unit: liters/hour
Arm/Group | Carfilzomib - Normal RF | Carfilzomib - Mild RI | Carfilzomib - Moderate RI | Carfilzomib - Severe RI | Carfilzomib - Dialysis
Number analyzed (Participants) | 0 | 0 | 1 | 1 | 0
liters/hour |  |  | 679 (NA) — Cannot be calculated for a sample of 1 | 46.6 (NA) — Cannot be calculated for a sample of 1 |

4. Secondary Outcome: Maximum Observed Plasma Concentration of Carfilzomib on Day 1 of Cycle 1
Time Frame: Cycle 1, Day 1, before dosing, at the end of the injection, 5, 15, 30, and 60 minutes, and 1.5, 2, 4, 6 and 24 hours postdose.
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Carfilzomib - Normal RF | Carfilzomib - Mild RI | Carfilzomib - Moderate RI | Carfilzomib - Severe RI | Carfilzomib - Dialysis
Number analyzed (Participants) | 8 | 9 | 5 | 5 | 8
ng/mL | 2077 (91.4) | 1623 (161) | 1840 (92.4) | 1231 (139) | 1539 (92.7)

5. Secondary Outcome: Maximum Observed Plasma Concentration of Carfilzomib on Day 15 of Cycle 1
Time Frame: as for outcome 2
Population: PK population with available data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Carfilzomib - Normal RF | Carfilzomib - Mild RI | Carfilzomib - Moderate RI | Carfilzomib - Severe RI | Carfilzomib - Dialysis
Number analyzed (Participants) | 7 | 8 | 5 | 4 | 6
ng/mL | 1768 (179) | 2406 (52.3) | 2627 (31.8) | 1914 (99.8) | 3236 (34.4)

6. Secondary Outcome: Maximum Observed Plasma Concentration of Carfilzomib on Day 15 of Cycle 2
Time Frame: Cycle 2, Day 15 before dosing, at the end of the injection, 5, 15, 30, and 60 minutes, and 1.5, 2, 4, 6 and 24 hours postdose.
Population: PK population with available data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Carfilzomib - Normal RF | Carfilzomib - Mild RI | Carfilzomib - Moderate RI | Carfilzomib - Severe RI | Carfilzomib - Dialysis
Number analyzed (Participants) | 0 | 0 | 1 | 2 | 0
ng/mL |  |  | 244 (NA) — Cannot be calculated for a sample of 1 | 3064 (3.9) |

7. Secondary Outcome: Area Under the Plasma Curve Extrapolated to Infinity (AUCinf) for Carfilzomib on Day 1 of Cycle 1
Time Frame: as for outcome 4
Population: PK evaluable population; AUCinf could not be estimated for 11 participants in the PK population who did not have adequate PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Carfilzomib - Normal RF | Carfilzomib - Mild RI | Carfilzomib - Moderate RI | Carfilzomib - Severe RI | Carfilzomib - Dialysis
Number analyzed (Participants) | 6 | 6 | 3 | 4 | 5
hr*ng/mL | 233 (51.6) | 241 (32.4) | 145 (111) | 172 (35.6) | 193 (55.2)

8. Secondary Outcome: Area Under the Plasma Curve Extrapolated to Infinity (AUCinf) for Carfilzomib on Day 15 of Cycle 1
Time Frame: as for outcome 2
Population: PK evaluable population with available data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Carfilzomib - Normal RF | Carfilzomib - Mild RI | Carfilzomib - Moderate RI | Carfilzomib - Severe RI | Carfilzomib - Dialysis
Number analyzed (Participants) | 5 | 5 | 3 | 1 | 5
hr*ng/mL | 127 (240) | 236 (44.3) | 257 (10.9) | 218 (NA) — Cannot be calculated for a sample of 1 | 272 (46.4)

9. Secondary Outcome: Area Under the Plasma Curve Extrapolated to Infinity (AUCinf) for Carfilzomib on Day 15 of Cycle 2
Time Frame: as for outcome 6
Population: PK evaluable population with available data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Carfilzomib - Normal RF | Carfilzomib - Mild RI | Carfilzomib - Moderate RI | Carfilzomib - Severe RI | Carfilzomib - Dialysis
Number analyzed (Participants) | 0 | 0 | 1 | 1 | 0
hr*ng/mL |  |  | 48.6 (NA) — Cannot be calculated for a sample of 1 | 579 (NA) — Cannot be calculated for a sample of 1 |

10. Secondary Outcome: Area Under the Concentration Time Curve to the Last Measurable Concentration (AUClast) for Carfilzomib on Day 1 of Cycle 1
Time Frame: as for outcome 1
Population: PK evaluable population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Carfilzomib - Normal RF | Carfilzomib - Mild RI | Carfilzomib - Moderate RI | Carfilzomib - Severe RI | Carfilzomib - Dialysis
Number analyzed (Participants) | 8 | 9 | 5 | 5 | 8
hr*ng/mL | 187 (75.3) | 194 (67.6) | 199 (91.3) | 135 (65.5) | 195 (65.3)

11. Secondary Outcome: Area Under the Concentration Time Curve to the Last Measurable Concentration (AUClast) for Carfilzomib on Day 15 of Cycle 1
Time Frame: as for outcome 2
Population: PK evaluable population with available data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Carfilzomib - Normal RF | Carfilzomib - Mild RI | Carfilzomib - Moderate RI | Carfilzomib - Severe RI | Carfilzomib - Dialysis
Number analyzed (Participants) | 7 | 8 | 5 | 4 | 6
hr*ng/mL | 159 (186) | 289 (58.5) | 371 (55.2) | 343 (53.1) | 264 (41.7)

12. Secondary Outcome: Area Under the Concentration Time Curve to the Last Measurable Concentration (AUClast) for Carfilzomib on Day 15 of Cycle 2
Time Frame: as for outcome 6
Population: PK evaluable population with available data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Carfilzomib - Normal RF | Carfilzomib - Mild RI | Carfilzomib - Moderate RI | Carfilzomib - Severe RI | Carfilzomib - Dialysis
Number analyzed (Participants) | 0 | 0 | 1 | 2 | 0
hr*ng/mL |  |  | 47.3 (NA) — Cannot be calculated for a sample of 1 | 345 (83.6) |

13. Secondary Outcome: Percentage of Carfilzomib Excreted Via Renal Elimination on Day 1 of Cycle 1
Description: The percentage of carfilzomib excreted in urine was calculated as the total amount excreted over 24 hours/dose.
Time Frame: Cycle 1, Day 1, 0-5 and 5-24 hours post-dose
Population: Participants in Groups 1-4 with available data
Measure: Mean (Standard Deviation); unit: percentage of carfilzomib dose
Arm/Group | Carfilzomib - Normal RF | Carfilzomib - Mild RI | Carfilzomib - Moderate RI | Carfilzomib - Severe RI | Carfilzomib - Dialysis
Number analyzed (Participants) | 8 | 8 | 7 | 5 | 0
percentage of carfilzomib dose | 0.490 (0.316) | 0.429 (0.271) | 0.160 (0.101) | 0.226 (0.0921) |

14. Secondary Outcome: Percentage of Carfilzomib Excreted Via Renal Elimination on Day 15 of Cycle 1
Description: The percentage of carfilzomib excreted in urine was calculated as the total amount excreted over 24 hours/dose.
Time Frame: Cycle 1, Day 15, 0-5 and 5-24 hours post-dose
Population: Participants in Groups 1-4 with available data
Measure: Mean (Standard Deviation); unit: percentage of carfilzomib dose
Arm/Group | Carfilzomib - Normal RF | Carfilzomib - Mild RI | Carfilzomib - Moderate RI | Carfilzomib - Severe RI | Carfilzomib - Dialysis
Number analyzed (Participants) | 7 | 6 | 5 | 4 | 0
percentage of carfilzomib dose | 0.446 (0.357) | 0.428 (0.262) | 0.202 (0.116) | 0.168 (0.0670) |

15. Secondary Outcome: Percentage of Carfilzomib Metabolites Excreted Via Renal Elimination on Day 1 of Cycle 1
Description: The percentage of the metabolites of carfilzomib (PR-389/M14 and PR-413/M15) excreted in urine was calculated as the total amount excreted over 24 hours/dose.
Time Frame: Cycle 1, Day 1, 0-5 and 5-24 hours post-dose
Population: Participants in Groups 1-4 with available data
Measure: Mean (Standard Deviation); unit: percentage of carfilzomib dose
Arm/Group | Carfilzomib - Normal RF | Carfilzomib - Mild RI | Carfilzomib - Moderate RI | Carfilzomib - Severe RI | Carfilzomib - Dialysis
Number analyzed (Participants) | 8 | 9 | 7 | 5 | 0
percentage of carfilzomib dose
  M14 | 33.1 (13.1) | 25.0 (4.81) | 21.7 (7.59) | 19.2 (4.36) |
  M15 | 1.93 (1.12) | 1.42 (0.314) | 0.776 (0.387) | 0.578 (0.230) |

16. Secondary Outcome: Percentage of Carfilzomib Metabolites Excreted Via Renal Elimination on Day 15 of Cycle 1
Description: as for outcome 15
Time Frame: Cycle 1, Day 15, 0-5 and 5-24 hours post-dose
Population: Participants in Groups 1-4 with available data
Measure: Mean (Standard Deviation); unit: percentage of carfilzomib dose
Arm/Group | Carfilzomib - Normal RF | Carfilzomib - Mild RI | Carfilzomib - Moderate RI | Carfilzomib - Severe RI | Carfilzomib - Dialysis
Number analyzed (Participants) | 7 | 6 | 5 | 4 | 0
percentage of carfilzomib dose
  M14 | 30.6 (11.6) | 27.0 (8.47) | 22.0 (6.89) | 17.0 (4.67) |
  M15 | 1.91 (1.03) | 1.55 (0.602) | 0.856 (0.377) | 0.475 (0.249) |

17. Secondary Outcome: Plasma Protein Binding (PPB) of Carfilzomib
Description: The plasma protein binding (PPB) of carfilzomib in plasma samples was determined using a rapid equilibrium dialysis (RED) device. Data are averages of the 3 time points (Cycle 1 Day 1, Cycle 1 Day 15, and Cycle 2 Day 15).
Time Frame: End of injection and 5 minutes post-dose on Cycle 1 Day 1, Cycle 1 Day 15, and Cycle 2 Day 15
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: percentage of carfilzomib bound
Arm/Group | Carfilzomib - Normal RF | Carfilzomib - Mild RI | Carfilzomib - Moderate RI | Carfilzomib - Severe RI | Carfilzomib - Dialysis
Number analyzed (Participants) | 11 | 8 | 9 | 9 | 7
percentage of carfilzomib bound
  End of Injection | 97.8 (0.6) | 97.6 (1.5) | 98.4 (0.4) | 98.2 (0.5) | 97.6 (0.7)
  5 minutes after injection | 98.1 (0.5) | 97.6 (1.6) | 98.2 (1.5) | 98.1 (0.8) | 98.2 (0.4)

18. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants with a best response of stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR) per the International Uniform Response Criteria for Multiple Myeloma.
  sCR: CR as defined below plus normal serum free light chain (sFLC) ratio and absence of clonal plasma cells in bone marrow by immunohistochemistry or immunofluorescence; CR: absence of M-protein in serum and urine confirmed by immunofixation and < 5% plasma cells in the bone marrow; VGPR: serum and urine M-proteins detectable by immunofixation, but not by electrophoresis or a ≥ 90% reduction in serum M-protein from baseline, plus a urine M-protein level of < 100 mg/24 hours; PR: reduction of M-protein in serum of ≥ 50% and in urine of ≥ 90% from baseline. If serum and urine M-protein were not measureable at baseline, a ≥ 50% decrease in the difference between involved and uninvolved sFLC levels from baseline.
Time Frame: From first dose until 30 days after the last dose; median duration of treatment across all groups was 121 days.
Population: The response evaluable population included all participants with measurable disease and a baseline and at least 1 post-baseline disease assessment or who discontinued study treatment due to a related adverse event prior to obtaining an on-study disease assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Carfilzomib - Normal RF | Carfilzomib - Mild RI | Carfilzomib - Moderate RI | Carfilzomib - Severe RI | Carfilzomib - Dialysis
Number analyzed (Participants) | 11 | 11 | 9 | 8 | 8
percentage of participants | 18.2 [2.3 to 51.8] | 27.3 [6.0 to 61.0] | 22.2 [2.8 to 60.0] | 25.0 [3.2 to 65.1] | 37.5 [8.5 to 75.5]

19. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Clinical benefit rate is defined as the percentage of participants whose best response was sCR, CR, VGPR, PR, or minimal response (MR), where MR is defined by the European Group for Blood and Marrow Transplant (EBMT) criteria as a reduction of M-protein in serum of 25% to 49% and in urine of 50% to 89% from baseline, maintained for at least 6 weeks.
Time Frame: From first dose until 30 days after the last dose; median duration of treatment across all groups was 121 days.
Population: The response evaluable population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Carfilzomib - Normal RF | Carfilzomib - Mild RI | Carfilzomib - Moderate RI | Carfilzomib - Severe RI | Carfilzomib - Dialysis
Number analyzed (Participants) | 11 | 11 | 9 | 8 | 8
percentage of participants | 27.3 [6.0 to 61.0] | 36.4 [10.9 to 69.2] | 22.2 [2.8 to 60.0] | 37.5 [8.5 to 75.5] | 37.5 [8.5 to 75.5]

20. Secondary Outcome: Duration of Response
Description: Duration of Response is defined as the time from first evidence of PR or better to confirmation of disease progression or death.
  Progressive disease was defined as any of the following:
  * An increase of more than 25% from nadir in any one of the following:
    * M-protein in serum (the absolute increase had to be ≥ 0.5 g/dL);
    * Urine (the absolute increase had to be ≥ 200 mg/24 hours);
    * The difference between involved and uninvolved sFLC (the absolute increase in the concentration of involved light chain had to be > 10 mg/dL);
    * ≥ 10% bone marrow infiltration by plasma cells;
  * Increased size of pre-existing bone lesions or plasmacytomas or new bone lesions or plasmacytomas.
  Median duration of response was estimated using the Kaplan-Meier method.
Time Frame: Participants were followed for disease progression for up to 2 years.
Population: Response Evaluable Population with a best overall response of sCR, CR, VGPR, or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carfilzomib - Normal RF | Carfilzomib - Mild RI | Carfilzomib - Moderate RI | Carfilzomib - Severe RI | Carfilzomib - Dialysis
Number analyzed (Participants) | 2 | 3 | 2 | 2 | 3
months | NA [2.0 to NA] — Could not be estimated due to the low number of events | NA [4.2 to NA] — Could not be estimated due to the low number of events | 14.8 [2.3 to 27.4] | NA [7.9 to NA] — Could not be estimated due to the low number of events | 7.9 [6.5 to 8.5]

21. Secondary Outcome: Time to Progression (TTP)
Description: Time to Progression is defined as the time from first dose of carfilzomib to disease progression. Median TTP was estimated using Kaplan-Meier methods.
Time Frame: Participants were followed for disease progression for up to 2 years.
Population: Response Evaluable Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carfilzomib - Normal RF | Carfilzomib - Mild RI | Carfilzomib - Moderate RI | Carfilzomib - Severe RI | Carfilzomib - Dialysis
Number analyzed (Participants) | 11 | 11 | 9 | 8 | 8
months | 4.4 [2.8 to 9.2] | 5.6 [0.5 to 7.9] | 2.8 [1.0 to 29.2] | 9.6 [1.0 to 11.8] | 6.5 [2.8 to 11.3]

ADVERSE EVENTS:
Time Frame: From the first dose of study drug until 30 days after the last dose. Median duration of treatment was 121 days.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Carfilzomib - Normal RF | Carfilzomib - Mild RI | Carfilzomib - Moderate RI | Carfilzomib - Severe RI | Carfilzomib - Dialysis
Serious Adverse Events (participants affected / at risk) | 5/12 | 8/12 | 10/10 | 6/8 | 8/8
Other Adverse Events (participants affected / at risk) | 12/12 | 12/12 | 10/10 | 8/8 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carfilzomib - Normal RF (N=12) | Carfilzomib - Mild RI (N=12) | Carfilzomib - Moderate RI (N=10) | Carfilzomib - Severe RI (N=8) | Carfilzomib - Dialysis (N=8)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 2 | 0
Right ventricular failure (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Disease progression (General disorders) | 0 | 3 | 0 | 1 | 3
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 1 | 0
Venoocclusive liver disease (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Amyloidosis (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Bronchitis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Central line infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 2 | 0 | 1
Injection site cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 2 | 4 | 2 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Respiratory tract infection bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 3 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 1 | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1 | 0 | 0
Superior vena caval occlusion (Vascular disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Carfilzomib - Normal RF (N=12) | Carfilzomib - Mild RI (N=12) | Carfilzomib - Moderate RI (N=10) | Carfilzomib - Severe RI (N=8) | Carfilzomib - Dialysis (N=8)
Anaemia (Blood and lymphatic system disorders) | 6 | 7 | 7 | 5 | 5
Hypocoagulable state (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 4 | 4 | 2 | 2 | 4
Neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 6 | 5 | 3 | 5
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 2
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 2
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Dilatation atrial (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 2 | 2 | 1
Ear congestion (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 1 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 1 | 0 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 2 | 0 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1
Bowel sounds abnormal (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Colonic haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 6 | 5 | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 5 | 6 | 5 | 2 | 4
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 6 | 4 | 6 | 1 | 4
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 3 | 0 | 3
Asthenia (General disorders) | 1 | 1 | 3 | 2 | 2
Catheter site haematoma (General disorders) | 0 | 0 | 1 | 0 | 0
Catheter site inflammation (General disorders) | 0 | 0 | 0 | 0 | 1
Catheter site related reaction (General disorders) | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 1 | 1 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 0 | 0 | 0
Chills (General disorders) | 1 | 2 | 1 | 0 | 0
Disease progression (General disorders) | 0 | 1 | 1 | 2 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 1
Facial pain (General disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 9 | 9 | 6 | 4 | 4
Generalised oedema (General disorders) | 0 | 0 | 1 | 0 | 0
Hypothermia (General disorders) | 0 | 0 | 0 | 0 | 1
Infusion related reaction (General disorders) | 1 | 0 | 0 | 0 | 0
Infusion site pain (General disorders) | 1 | 0 | 0 | 1 | 1
Local swelling (General disorders) | 1 | 0 | 1 | 0 | 0
Mass (General disorders) | 0 | 1 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0
Oedema (General disorders) | 2 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 4 | 2 | 3 | 3 | 1
Pain (General disorders) | 0 | 3 | 4 | 0 | 4
Pitting oedema (General disorders) | 1 | 0 | 1 | 1 | 0
Pyrexia (General disorders) | 3 | 2 | 3 | 0 | 4
Tenderness (General disorders) | 0 | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Paronychia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 1 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 3
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 1 | 3 | 2
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Post procedural vomiting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Postoperative fever (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Abdominal bruit (Investigations) | 1 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 2 | 0 | 2
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0 | 0 | 1
Blood albumin decreased (Investigations) | 0 | 1 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood calcium increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood creatinine decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 2 | 5 | 1 | 2
Blood glucose decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood phosphorus decreased (Investigations) | 1 | 0 | 2 | 0 | 1
Blood phosphorus increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood potassium decreased (Investigations) | 3 | 0 | 1 | 0 | 2
Blood potassium increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood pressure diastolic decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 1 | 1 | 0 | 0 | 0
Blood sodium decreased (Investigations) | 0 | 2 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 2 | 3 | 1 | 3
Breath sounds abnormal (Investigations) | 0 | 2 | 3 | 1 | 0
Carbon dioxide decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Cardiac murmur (Investigations) | 0 | 2 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 1 | 1 | 1
International normalised ratio increased (Investigations) | 1 | 0 | 1 | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 1 | 0 | 0 | 2
Occult blood positive (Investigations) | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 1 | 0 | 1 | 0 | 1
Respiratory rate decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 1
Urine output decreased (Investigations) | 0 | 0 | 2 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 1 | 2 | 2 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 2
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 3 | 4 | 2 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 4 | 4 | 2 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Overweight (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 3 | 1 | 1 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2 | 2 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1 | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1
Nodule on extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 1 | 0 | 1 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 3
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Shoulder pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0 | 1
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Areflexia (Nervous system disorders) | 1 | 2 | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Diplegia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 2 | 2 | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 5 | 2 | 2 | 0 | 2
Hypoaesthesia (Nervous system disorders) | 2 | 3 | 1 | 2 | 1
Hyporeflexia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Neuropathic pain (Nervous system disorders) | 3 | 4 | 0 | 0 | 2
Neuropathy (Nervous system disorders) | 1 | 0 | 0 | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 2 | 1 | 2 | 2 | 0
Paraesthesia (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 1 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 2 | 1 | 1 | 0 | 2
Insomnia (Psychiatric disorders) | 3 | 1 | 2 | 2 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Azotaemia (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0
Incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Urine flow decreased (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 4 | 3 | 3
Dyspnoea exacerbated (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Blood blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin tightness (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 2 | 1 | 2
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 4
Pallor (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Superior vena caval occlusion (Vascular disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.